CLINICAL TRIAL: NCT01023035
Title: Boceprevir and Peginterferon/Ribavirin for the Treatment of Chronic Hepatitis C in Treatment-Naive Subjects: A Comparison of Erythropoietin Use Versus Ribavirin Dose Reduction for the Management of Anemia
Brief Title: Boceprevir/Peginterferon/Ribavirin for Chronic Hepatitis C: Erythropoietin Use Versus Ribavirin Dose Reduction for Anemia (P06086 AM2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06086; 2009-012782-63 (EudraCT Number)
Record Dates: First submitted 2009-11-24; First posted 2009-12-01 (Estimated); Results first posted 2012-11-15 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin; Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treated/Not Randomized (Experimental): Participants received 4 weeks of PEG2b/RBV followed by 24 or 44 weeks of boceprevir plus PEG2b/RBV depending on Hepatitis C Virus RNA (HCV-RNA) levels. Participants continued with this treatment if their serum hemoglobin remained >10 g/dL throughout the 28- or 48-week treatment period.
  Interventions: Drug: Boceprevir; Drug: Peginterferon alfa-2b (PEG2b); Drug: Ribavirin (RBV)
- Ribavirin Dose Reduction (Experimental): After the initiation of treatment with 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin = ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Ribavirin (RBV) Dose Reduction Arm received reduced doses of RBV for management of the anemia in combination with PEG2b and boceprevir therapies.
  Interventions: Drug: Boceprevir; Drug: Peginterferon alfa-2b (PEG2b); Drug: Ribavirin (RBV)
- Erythropoietin Use (Experimental): After the initiation of treatment with 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin = ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Erythropoietin Use Arm received erythropoietin for management of the anemia in addition to PEG2b/RBV and boceprevir therapies.
  Interventions: Drug: Boceprevir; Drug: Peginterferon alfa-2b (PEG2b); Drug: Ribavirin (RBV); Drug: Erythropoietin

INTERVENTIONS:
Drug: Boceprevir — 800 mg given three times a day (TID), orally (PO)
  Other Names: SCH 503034
Drug: Peginterferon alfa-2b (PEG2b) — 1.5 µg/kg/week given subcutaneously (SC)
  Other Names: SCH 054031
Drug: Ribavirin (RBV) — Ribavirin weight-based dosing (WBD), 600 to 1400 mg/day given twice daily (BID), orally (PO)
  Other Names: SCH 018908, Rebetol
Drug: Erythropoietin — Initial dose of 40,000 Units given subcutaneously (SC) once weekly (QW), with dose adjustment as necessary to achieve and maintain serum hemoglobin levels of 10-12 g/dL
  Other Names: Procrit, Eprex
  Arms: Erythropoietin Use

SUMMARY:
The current trial is designed to prospectively explore the safety of erythropoietin use for the treatment of anemia during boceprevir plus peginterferon alfa-2b/Ribavirin (PEG2b/RBV) therapy and to assess its relationship to efficacy. All participants in this trial will be treated with the triple combination of boceprevir plus PEG2b/RBV. If a participant becomes anemic during treatment, the participant will be randomized to one of two therapeutic strategies for management of anemia (erythropoietin use versus RBV dose reduction).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have previously documented Chronic Hepatitis C (CHC) genotype 1 infection.
* Hemoglobin concentration at Screening must be ≤15 g/dL for both females and males.
* Participant must have a liver biopsy with histology consistent with CHC and no other etiology.
* Participant with bridging fibrosis (F3) or cirrhosis (F4) must have an ultrasound within 6 months of the Screening Visit (or between Screening and Day 1) with no findings suspicious for hepatocellular carcinoma.
* Participant's weight must be ≥40 kg and ≤125 kg.
* Participant and participant's partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study medication, or longer if dictated by local regulations.
* Participant must be willing to give written informed consent.
* Participant must be willing to attend frequent site visits for the duration of the trial.
* Participant must not have any contraindications for the use of erythropoietin.

Exclusion Criteria:

* Participants known to be coinfected with the human immunodeficiency virus (HIV) or hepatitis B virus.
* Participants who received prior treatment for hepatitis C.
* Treatment with any investigational drug within 30 days of the screening visit in this trial.
* Participants receiving any of the following medication(s) within 2 weeks prior to the Day 1 visit: alfuzosin, antiarrhythmics (amiodarone, bepridil, flecainide, propafenone, and quinidine), ergot derivatives, cisapride, lovastatin, simvastatin, pimozide, triazolam, and orally administered midazolam.
* Participation in any other clinical trial within 30 days of the screening visit in this trial or intention to participate in another clinical trial during participation in this trial.
* Evidence of decompensated liver disease.
* Diabetic and/or hypertensive participants with clinically significant ocular examination findings.
* Pre-existing psychiatric condition(s).
* Clinical diagnosis of substance abuse of specified drugs within specified timeframes.
* Any known pre-existing medical condition that could interfere with the participant's participation in and completion of the trial.
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin).
* Participants who are pregnant or nursing. Participants who intend to become pregnant during the trial period. Male participants with partners who are, or intend to become, pregnant during the trial period.
* Any other condition which, in the opinion of a physician, would make the participant unsuitable for enrollment or could interfere with the participant participating in and completing the trial.
* Participant who had a life-threatening serious adverse event during the screening period.
* A participant must not be a member or a family member of the personnel of the investigational or sponsor staff directly involved with this trial.
* Protocol-specified hematologic, biochemical, and serologic criteria (growth factors may not be used to achieve trial entry requirements).
* Serum albumin below the lower limit of normal (LLN) of laboratory reference range.
* Thyroid-stimulating hormone (TSH) >1.2 x Upper Limit of Normal (ULN) or <0.8 x LLN of laboratory reference.
* Serum creatinine >ULN of the laboratory reference.
* Protocol-specified serum glucose concentrations.
* Prothrombin time/partial thromboplastin time (PT/PTT) values >10% above laboratory reference range.
* Protocol-specified alpha fetoprotein concentrations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2009-12-07 (Actual); Primary Completion 2011-10-26 (Actual); Study Completion 2011-10-26 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Poordad F, Lawitz E, Reddy KR, Afdhal NH, Hezode C, Zeuzem S, Lee SS, Calleja JL, Brown RS Jr, Craxi A, Wedemeyer H, Nyberg L, Nelson DR, Rossaro L, Balart L, Morgan TR, Bacon BR, Flamm SL, Kowdley KV, Deng W, Koury KJ, Pedicone LD, Dutko FJ, Burroughs MH, Alves K, Wahl J, Brass CA, Albrecht JK, Sulkowski MS; Protocol 6086 Investigators. Effects of ribavirin dose reduction vs erythropoietin for boceprevir-related anemia in patients with chronic hepatitis C virus genotype 1 infection--a randomized trial. Gastroenterology. 2013 Nov;145(5):1035-1044.e5. doi: 10.1053/j.gastro.2013.07.051. Epub 2013 Aug 4. PMID 23924660

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 687 Participants enrolled and were treated with Peginterferon/Ribavirin (PEG2b/RBV) followed by PEG2b/RBV + boceprevir. 500 participants became anemic during treatment and were randomized to either the RBV Dose Reduction Arm (n=249) or the Erythropoietin Use Arm (n=251).
Groups:
- Ribavirin Dose Reduction Arm: After the initiation of treatment with 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin = ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Ribavirin (RBV) Dose Reduction Arm received reduced doses of RBV for management of the anemia in combination with PEG2b and boceprevir therapies.
- Erythropoietin Use Arm: After the initiation of treatment with 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin = ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Erythropoietin Use Arm received erythropoietin for management of the anemia in addition to PEG2b/RBV and boceprevir therapies.
Period: Treatment Period
Arm/Group | Ribavirin Dose Reduction Arm | Erythropoietin Use Arm | Treated/Not Randomized
Started | 249 | 251 | 187
Completed | 177 | 166 | 69
Not Completed | 72 | 85 | 118
Not completed — Adverse Event | 27 | 32 | 50
Not completed — Non-Medical Reasons | 19 | 22 | 44
Not completed — Treatment Failure | 26 | 31 | 24
Period: Follow-up Period (up to Week 72)
Arm/Group | Ribavirin Dose Reduction Arm | Erythropoietin Use Arm | Treated/Not Randomized
Started | 238 | 235 | 147
Completed | 210 | 207 | 108
Not Completed | 28 | 28 | 39
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Non-medical Reason | 26 | 28 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribavirin Dose Reduction Arm | Erythropoietin Use Arm | Treated/Not Randomized | Total
Number analyzed (Participants) | 249 | 251 | 187 | 687
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.9) | 49.7 (9.7) | 47.5 (10.1) | 49.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 164 | 99 | 434
  Male | 78 | 87 | 88 | 253

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR)
Description: SVR was defined as undetectable plasma Hepatitis C Virus ribonucleic acid (HCV-RNA) at Follow-up Week 24
Time Frame: At Follow-up Week 24
Population: The primary efficacy analysis was performed on all participants who were randomized to either the RBV Dose Reduction Arm or the EPO Use Arm for anemia management (i.e. the Full Analysis Set of patients requiring anemia management [FAS, n=500]).
Measure: Number; unit: percentage of participants
Groups:
- Ribavirin Dose Reduction Arm: After treatment for 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin of ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Ribavirin (RBV) Dose Reduction Arm received reduced doses of RBV for management of the anemia in combination with PEG2b and boceprevir therapies.
- Erythropoietin Use Arm: After treatment for 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin of ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Erythropoietin Use Arm received erythropoietin for management of the anemia in addition to PEG2b/RBV and boceprevir therapies.
Arm/Group | Ribavirin Dose Reduction Arm | Erythropoietin Use Arm
Number analyzed (Participants) | 249 | 251
percentage of participants | 71.5 | 70.9
Statistical Analysis 1: Comparison: Ribavirin Dose Reduction Arm vs Erythropoietin Use Arm; The modified Koch method was used to calculate the stratum-adjusted Mantel-Haenszel (MH) difference between the SVR rates for the Erythropoietin Use Arm versus the Ribavirin Dose Reduction Arm and corresponding 95% confidence interval with continuity correction; Test type: Superiority or Other; Mantel-Haenszel, modified Koch method; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-8.6 to 7.2]

2. Secondary Outcome: Percentage of Participants Who Discontinued Treatment
Description: Cumulative discontinuation was defined as the sum of discontinuations due to adverse events, viral breakthrough/resistance, detectable HCV-RNA and futility rules (<2-log10 decline in HCV-RNA at Treatment Week 12, ≥ Lower Limit of Quantification [LLQ] HCV-RNA at Treatment Week 24), and other (noncompliance, withdrawal of consent, lost to follow-up).
Time Frame: From Study Day 1 up to Study Treatment Week 48
Population: All Treated Participants, defined as all participants who were treated with any study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ribavirin Dose Reduction Arm: After treatment for 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin = ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Ribavirin (RBV) Dose Reduction Arm received reduced doses of RBV for management of the anemia in combination with PEG2b and boceprevir therapies.
- Erythropoietin Use Arm: After treatment for 4 weeks with PEG2b/RBV followed by 24 or 44 weeks of boceprevir, participants who became anemic (serum hemoglobin = ≤10 g/dL) within the 28- or 48-week treatment period and who were randomized to the Erythropoietin Use Arm received erythropoietin for management of the anemia in addition to PEG2b/RBV and boceprevir therapies.
Arm/Group | Ribavirin Dose Reduction Arm | Erythropoietin Use Arm | Treated/Not Randomized
Number analyzed (Participants) | 249 | 251 | 187
percentage of participants | 29 [23 to 35] | 34 [28 to 40] | 63 [56 to 70]

ADVERSE EVENTS:
Arm/Group | Ribavirin Dose Reduction Arm | Erythropoietin Use Arm | Treated/Not Randomized
Serious Adverse Events (participants affected / at risk) | 39/249 | 33/251 | 15/187
Other Adverse Events (participants affected / at risk) | 247/249 | 248/251 | 180/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ribavirin Dose Reduction Arm (N=249) | Erythropoietin Use Arm (N=251) | Treated/Not Randomized (N=187)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 7 (7) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden Cardiac Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis Obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess Soft Tissue (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corneal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Tubo-ovarian Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple Drug Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Operative Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Snake Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood Potassium Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 0 (0)
Diabetes Melllitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Arthraliga (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VIIth Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal Behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adnexa Uteri Mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosed Varicose Vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ribavirin Dose Reduction Arm (N=249) | Erythropoietin Use Arm (N=251) | Treated/Not Randomized (N=187)
Anaemia (Blood and lymphatic system disorders) | 172 (239) | 152 (215) | 8 (10)
Leukopenia (Blood and lymphatic system disorders) | 18 (29) | 21 (54) | 8 (10)
Neutropenia (Blood and lymphatic system disorders) | 71 (154) | 81 (162) | 30 (49)
Hypothyroidism (Endocrine disorders) | 15 (16) | 11 (11) | 5 (5)
Vision Blurred (Eye disorders) | 18 (19) | 14 (14) | 12 (12)
Abdominal Pain (Gastrointestinal disorders) | 20 (23) | 16 (18) | 10 (15)
Abdominal Pain Upper (Gastrointestinal disorders) | 16 (18) | 12 (13) | 7 (7)
Constipation (Gastrointestinal disorders) | 16 (16) | 22 (23) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 77 (102) | 87 (107) | 52 (70)
Dry Mouth (Gastrointestinal disorders) | 16 (17) | 30 (30) | 17 (17)
Dysguesia (Gastrointestinal disorders) | 85 (94) | 100 (104) | 61 (67)
Dyspepsia (Gastrointestinal disorders) | 16 (16) | 24 (33) | 9 (11)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 20 (21) | 13 (13) | 14 (16)
Mouth Ulceration (Gastrointestinal disorders) | 3 (3) | 14 (14) | 4 (4)
Nausea (Gastrointestinal disorders) | 127 (171) | 153 (211) | 94 (118)
Stomatitis (Gastrointestinal disorders) | 19 (20) | 20 (22) | 10 (11)
Vomiting (Gastrointestinal disorders) | 49 (66) | 62 (103) | 38 (48)
Asthenia (General disorders) | 21 (32) | 19 (29) | 16 (22)
Chills (General disorders) | 72 (78) | 79 (86) | 49 (54)
Fatigue (General disorders) | 174 (237) | 178 (248) | 108 (138)
Influenza Like Illness (General disorders) | 68 (74) | 67 (75) | 44 (47)
Injection Site Erythema (General disorders) | 27 (28) | 33 (37) | 21 (21)
Injection Site Reaction (General disorders) | 23 (25) | 36 (36) | 21 (25)
Irritability (General disorders) | 51 (62) | 64 (74) | 41 (44)
Oedema Peripheral (General disorders) | 17 (19) | 6 (6) | 5 (7)
Pain (General disorders) | 19 (21) | 37 (43) | 21 (22)
Pyrexia (General disorders) | 55 (63) | 70 (114) | 45 (52)
Bronchitis (Infections and infestations) | 9 (9) | 13 (14) | 6 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 13 (13) | 12 (14) | 10 (10)
Urinary Tract Infection (Infections and infestations) | 14 (22) | 8 (9) | 9 (9)
Weight Decreased (Investigations) | 19 (20) | 39 (53) | 22 (26)
Decreased Appetite (Metabolism and nutrition disorders) | 61 (65) | 65 (71) | 51 (56)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (55) | 58 (68) | 34 (41)
Back Pain (Musculoskeletal and connective tissue disorders) | 31 (33) | 19 (20) | 15 (19)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 (11) | 12 (16) | 11 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 56 (64) | 60 (66) | 28 (36)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 13 (15) | 8 (10)
Disturbance in Attention (Nervous system disorders) | 21 (23) | 42 (46) | 20 (24)
Dizziness (Nervous system disorders) | 58 (70) | 67 (85) | 37 (38)
Headache (Nervous system disorders) | 119 (151) | 136 (168) | 77 (92)
Hypoaesthesia (Nervous system disorders) | 14 (20) | 11 (14) | 4 (4)
Paraesthesia (Nervous system disorders) | 16 (17) | 14 (17) | 11 (15)
Affect Lability (Psychiatric disorders) | 10 (11) | 14 (14) | 9 (11)
Anxiety (Psychiatric disorders) | 29 (33) | 30 (36) | 28 (31)
Depression (Psychiatric disorders) | 50 (60) | 52 (65) | 38 (41)
Insomnia (Psychiatric disorders) | 72 (81) | 75 (89) | 60 (63)
Cough (Respiratory, thoracic and mediastinal disorders) | 57 (65) | 61 (71) | 32 (42)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 (55) | 52 (60) | 26 (30)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 26 (32) | 29 (35) | 16 (20)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 26 (31) | 9 (9)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 17 (21) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 95 (102) | 99 (108) | 55 (57)
Dry Skin (Skin and subcutaneous tissue disorders) | 45 (47) | 44 (45) | 21 (22)
Pruritis (Skin and subcutaneous tissue disorders) | 44 (56) | 57 (68) | 21 (31)
Rash (Skin and subcutaneous tissue disorders) | 70 (94) | 61 (100) | 34 (40)
Rash Generalised (Skin and subcutaneous tissue disorders) | 4 (4) | 13 (13) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts.